CLINICAL TRIAL: NCT02488642
Title: Medical Management of Late Intrauterine Death Using a Therapeutic Combination of Isosorbide Dinitrate and Oxytocin.
Brief Title: Medical Management of Late Intrauterine Death.
Acronym: INPer
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute of Perinatology (Other Government)
Collaborators: National Council of Science and Technology, Mexico (Other)
Responsible Party: Principal Investigator, Gabriel Arteaga Troncoso, Medical Researcher, National Institute of Perinatology
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 212250-29021
Record Dates: First submitted 2015-06-26; First posted 2015-07-02 (Estimated); Last update posted 2015-07-24 (Estimated); Status verified 2015-07

CONDITIONS: Cervical Pregnancy; Maternal Care for Late Fetal Death
Keywords: Isosorbide dinitrate gel solution; late intrauterine death; nitric oxide donors
MeSH Terms: interventions — Isosorbide Dinitrate; Isosorbide; Misoprostol; Oxytocin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- isosorbide dinitrate-oxytocin (Experimental): Preinduction with isosorbide dinitrate gel solution (80 mg/1.5 mL) were administered in the posterior fornix every 3 hours. Once a Bishop score of over 7 was reached, oxytocin was infused in a balanced electrolyte solution beginning with an infusion rate of 2 milli-International Units per minute (mIU/min) and doubling the dose every 15 minutes.
  If the cervical conditions (<7 Bishop Score) did not change after the treatment application, a new dose, without exceeding 4 doses, to facilitate cervical ripening.
  Interventions: Drug: Isosorbide Dinitrate; Drug: Oxytocin
- misoprostol-oxytocin (Placebo Comparator): Preinduction with misoprostol gel solution (100 mcg/1.5 mL) were administered in the posterior fornix every 3 hours. Once a Bishop score of over 7 was reached, oxytocin was infused in a balanced electrolyte solution beginning with an infusion rate of 2 milli-International Units per minute (mIU/min) and doubling the dose every 15 minutes.
  If the cervical conditions (<7 Bishop score) did not change after the treatment application, participants received a new dose, without exceeding 4 doses, to facilitate cervical ripening.
  Interventions: Drug: Misoprostol; Drug: Oxytocin

INTERVENTIONS:
Drug: Isosorbide Dinitrate
  Other Names: Isordil; Dilatrate-SR; Sorbitrate
  Arms: isosorbide dinitrate-oxytocin
Drug: Misoprostol
  Other Names: Cytotec
  Arms: misoprostol-oxytocin
Drug: Oxytocin — Oxytocin was infused in a balanced electrolyte solution beginning with an infusion rate of 2 milli-International Units per minute (mIU/min) and doubling the dose every 15 minutes.

SUMMARY:
The purpose of this study is to assess the therapeutic efficacy and safety of isosorbide dinitrate-oxytocin in combination in the management of late intrauterine foetal death.

DETAILED DESCRIPTION:
A prospective, randomised, double-blind, controlled clinical trial (RCT) was conducted to compare the efficacy and clinical safety of the induction of labour using the combination of isosorbide dinitrate-oxytocin (experimental arm, X = 1) compared to misoprostol-oxytocin (standard arm, X = 0). The main result of the study was the success rate of foetal expulsion within 15 hours, while the average administration induction interval defined the secondary result. A total of 60 women with pregnancies greater than 20 weeks gestation were referred for foetal evacuation. We defined late intrauterine foetal death (IUFD) as babies without signs of life in the uterus after 20 complete weeks of pregnancy. The approval to conduct the study was obtained from the institutional board ethical committees of both hospitals. All participants were informed about the objectives of the study, and informed consent was required. Patients with the following characteristics were included: closed cervix without evidence of cervical dilation or baseline uterine activity, A Bishop score of <5, having intact membranes, gestation greater than or equal to 20 weeks established by the date of menstruation or by fetometry and ultrasound-confirmed late IUFD. This study did not include the medical management of multiple pregnancies, IUFD after late foeticide or the management of specific medical conditions associated with an increase in the risk of IUFD or patients with a history of hypertension, along with women with a history of unexplained antepartum haemorrhage, pelvic dystocia or any another counter-indications where medications were used. Patients were assigned through a computational random number generator to receive isosorbide dinitrate or misoprostol. Allocation to groups was predetermined and arranged in numerical order. All participants were given a vaginal exam by the same person, who was blinded to the treatment allocation. The medications were administered in the posterior fornix, and cervical activity was evaluated at baseline and every 3 hours to monitor any change based on the Bishop score.

If the cervical conditions did not change after the treatment application, participants received a new dose, without exceeding 4 doses, to facilitate cervical ripening. Once a Bishop score of over 7 was reached, oxytocin was infused in a balanced electrolyte solution beginning with an infusion rate of 2 milli-International Units per minute (mIU/min) and doubling the dose every 15 minutes. The labour induction time from the first application of medication to the expulsion of the foetus was determined with a digital stopwatch. Each woman's vital signs were verified to determine that she was in stable condition and demonstrated haemodynamic stability as a requirement for the application of a new dose. During this time, the data and medical information were collected on paper and were later entered into a computational database. The participants remained at rest during the evaluation of adverse effects, such as headache, abdominal pain, pelvic pain, lower back pain, nausea, dizziness, and vomiting. The lack of cervical activity after 4 doses of medication was considered treatment failure.

A base solution of isosorbide dinitrate and misoprostol was prepared to obtain a concentration of 20 micrograms per milliliter (mcg/mL) in 10% lactose solution. Serial dilutions were performed using known concentrations in mobile phase buffer solution (150 g ammonium acetate and 11.5 mL glacial acetic acid to 1 L water), methanol and water in a proportion of 350:100:550, respectively. The concentration of both drugs was determined using a ultraviolet (UV) light spectrophotometer reading at lambda 220 nm and a reference filter of lambda 278 nm. The mean absorbance for each set of standards, controls and samples was calculated by a standard plot curve. Computer-based curve-fitting statistical software was employed. Peak absorption and area under the curve were taken into account to determine stability of the pharmacological integration. Known samples of isosorbide dinitrate and misoprostol were added to 100% glycerin to prepare the gel solution. The reagents had final concentrations of either 80 mg of isosorbide dinitrate in 1.5 ml of gel solution or 100 micrograms of misoprostol in the same presentation.

Both solutions were packed in syringes that had the same appearance for the purpose of keeping the physician, patient and researcher blinded. The pharmacist was the only participant who knew the contents of the syringes. Four syringes were placed in an opaque and sealed envelope consecutively numbered with a unique study number. The envelopes were opened by the physician who applied the contents of the syringe, repeating the administration every 3 hours according to the prior selection and random allocation of patients. The entire "stock" of reagents remained stable for a period of 20 days and was maintained at room temperature (18-25° C) before using.

The calculation of the sample size was based on the Cox regression model using the risk quotient (log Hazard Ratio) and a 95% confidence interval (95% CI).17 To reach a power (superiority of the clinical trial) of 80% and an α value of 0.05, with a standard deviation of 0.5 and under the assumption that 25% of all women will fail to induce labour, the estimated sample size required for the trial was 60 patients (30 in each arm).

All continuous variables were summarised using histograms and the measures of central tendency before conducting the statistical analyses. The statistical analyses were performed using the Chi-Square test, Fisher's exact test and the Mantel-Haenszel test, and Student's t test when appropriate. The Shapiro-Wilk test was used to verify the normality of the data. To model the time-event of labour induction after IUFD, Cox regression was utilised, controlling for the covariates maternal age, foetal size and weight, and weeks of gestation. The proportional hazards assumption was evaluated using the two graphed lines, which corresponded to the survival curves (absence of crossing) and the log-log plots in the figure. Respiratory and cardiac rate, temperature (measured orally) and systolic and diastolic blood pressures (recorded using sphygmomanometry) were determined at baseline and every 3 hours until the trial ended. Relative risks (RRs) and 95% CIs were estimated utilising bivariate analysis, including non-serious adverse events among the treatment groups. Attributable risk was calculated to determine the probability of total risk of each adverse effect observed with the use of isosorbide dinitrate or misoprostol. All of the tests were two-tailed, and results that had values of p < 0.05 were considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Closed cervix without evidence of cervical dilation or baseline uterine activity.
* A Bishop score of <5, having intact membranes.
* Gestation greater than or equal to 20 weeks established by the date of menstruation or by fetometry and ultrasound-confirmed late IUFD.

Exclusion Criteria:

* Multiple pregnancies.
* IUFD after late foeticide or the management of specific medical conditions associated with an increase in the risk of IUFD.
* Patients with a history of hypertension.
* Women with a history of unexplained antepartum haemorrhage, pelvic dystocia or any another counter-indications where medications were used.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-05; Primary Completion 2013-09 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Rates of uterine expulsion in the women who received the isosorbide dinitrate-oxytocin regimen | within 15 hours of administration

SECONDARY OUTCOMES:
A Bishop score of >7 of administration of the first dose of isosorbide dinitrate | within 12 hours

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel Arteaga-Troncoso, PhD., Principal Investigator — National Institute of Perinatology

REFERENCES:
- [Background] World Health Organization. Induction and augmentation of labour. In: WHO, UNFPA, UNICEF, World Bank, editor. Managing Complications in Pregnancy and Childbirth: A Guide for Midwives and Doctors. Geneva: WHO; 2000. pp. 17-25.
- [Result] Koopmans L, Wilson T, Cacciatore J, Flenady V. Support for mothers, fathers and families after perinatal death. Cochrane Database Syst Rev. 2013 Jun 19;2013(6):CD000452. doi: 10.1002/14651858.CD000452.pub3. PMID 23784865
- [Result] Radestad I, Steineck G, Nordin C, Sjogren B. Psychological complications after stillbirth--influence of memories and immediate management: population based study. BMJ. 1996 Jun 15;312(7045):1505-8. doi: 10.1136/bmj.312.7045.1505. PMID 8646141
- [Result] Silver RM, Heuser CC. Stillbirth workup and delivery management. Clin Obstet Gynecol. 2010 Sep;53(3):681-90. doi: 10.1097/GRF.0b013e3181eb3297. PMID 20661052
- [Result] Hughes EG, Kelly AJ, Kavanagh J. Dinoprostone vaginal insert for cervical ripening and labor induction: a meta-analysis. Obstet Gynecol. 2001 May;97(5 Pt 2):847-55. doi: 10.1016/s0029-7844(00)01216-3. PMID 11336776
- [Result] Neiger R, Greaves PC. Comparison between vaginal misoprostol and cervical dinoprostone for cervical ripening and labor induction. Tenn Med. 2001 Jan;94(1):25-7. PMID 11194687
- [Result] Bolnick JM, Velazquez MD, Gonzalez JL, Rappaport VJ, McIlwain-Dunivan G, Rayburn WF. Randomized trial between two active labor management protocols in the presence of an unfavorable cervix. Am J Obstet Gynecol. 2004 Jan;190(1):124-8. doi: 10.1016/s0002-9378(03)00952-9. PMID 14749647
- [Result] Khan RU, El-Refaey H, Sharma S, Sooranna D, Stafford M. Oral, rectal, and vaginal pharmacokinetics of misoprostol. Obstet Gynecol. 2004 May;103(5 Pt 1):866-70. doi: 10.1097/01.AOG.0000124783.38974.53. PMID 15121558
- [Result] Arteaga-Troncoso G, Villegas-Alvarado A, Belmont-Gomez A, Martinez-Herrera FJ, Villagrana-Zesati R, Guerra-Infante F. Intracervical application of the nitric oxide donor isosorbide dinitrate for induction of cervical ripening: a randomised controlled trial to determine clinical efficacy and safety prior to first trimester surgical evacuation of retained products of conception. BJOG. 2005 Dec;112(12):1615-9. doi: 10.1111/j.1471-0528.2005.00760.x. PMID 16305563
- [Result] Ignarro LJ, Lippton H, Edwards JC, Baricos WH, Hyman AL, Kadowitz PJ, Gruetter CA. Mechanism of vascular smooth muscle relaxation by organic nitrates, nitrites, nitroprusside and nitric oxide: evidence for the involvement of S-nitrosothiols as active intermediates. J Pharmacol Exp Ther. 1981 Sep;218(3):739-49. No abstract available. PMID 6115052
- [Result] Ignarro LJ. Heme-dependent activation of soluble guanylate cyclase by nitric oxide: regulation of enzyme activity by porphyrins and metalloporphyrins. Semin Hematol. 1989 Jan;26(1):63-76. No abstract available. PMID 2564216
- [Result] Schmidt HH, Lohmann SM, Walter U. The nitric oxide and cGMP signal transduction system: regulation and mechanism of action. Biochim Biophys Acta. 1993 Aug 18;1178(2):153-75. doi: 10.1016/0167-4889(93)90006-b. No abstract available. PMID 7688574
- [Result] Murad F. Regulation of cytosolic guanylyl cyclase by nitric oxide: the NO-cyclic GMP signal transduction system. Adv Pharmacol. 1994;26:19-33. doi: 10.1016/s1054-3589(08)60049-6. PMID 7913616
- [Result] Chung SJ, Fung HL. Identification of the subcellular site for nitroglycerin metabolism to nitric oxide in bovine coronary smooth muscle cells. J Pharmacol Exp Ther. 1990 May;253(2):614-9. PMID 2110975
- [Result] Feelisch M, Kelm M. Biotransformation of organic nitrates to nitric oxide by vascular smooth muscle and endothelial cells. Biochem Biophys Res Commun. 1991 Oct 15;180(1):286-93. doi: 10.1016/s0006-291x(05)81290-2. PMID 1656970
- [Result] Michel T, Smith TW. Nitric oxide synthases and cardiovascular signaling. Am J Cardiol. 1993 Sep 9;72(8):33C-38C. doi: 10.1016/0002-9149(93)90253-9. PMID 7690516
- [Result] Hsieh FY, Lavori PW. Sample-size calculations for the Cox proportional hazards regression model with nonbinary covariates. Control Clin Trials. 2000 Dec;21(6):552-60. doi: 10.1016/s0197-2456(00)00104-5. PMID 11146149
- [Result] Wagaarachchi PT, Ashok PW, Narvekar NN, Smith NC, Templeton A. Medical management of late intrauterine death using a combination of mifepristone and misoprostol. BJOG. 2002 Apr;109(4):443-7. doi: 10.1111/j.1471-0528.2002.01238.x. PMID 12013166
- [Result] Espey MG, Miranda KM, Feelisch M, Fukuto J, Grisham MB, Vitek MP, Wink DA. Mechanisms of cell death governed by the balance between nitrosative and oxidative stress. Ann N Y Acad Sci. 2000;899:209-21. doi: 10.1111/j.1749-6632.2000.tb06188.x. PMID 10863541
- [Result] Rapoport RM, Draznin MB, Murad F. Endothelium-dependent vasodilator-and nitrovasodilator-induced relaxation may be mediated through cyclic GMP formation and cyclic GMP-dependent protein phosphorylation. Trans Assoc Am Physicians. 1983;96:19-30. No abstract available. PMID 6149646
- [Result] Lokugamage AU, Forsyth SF, Sullivan KR, El Refaey H, Rodeck CH. Randomized trial in multiparous patients: investigating a single vs. two-dose regimen of intravaginal misoprostol for induction of labor. Acta Obstet Gynecol Scand. 2003 Feb;82(2):138-42. doi: 10.1034/j.1600-0412.2003.00084.x. PMID 12648175
- [Result] Cabrol D, Dubois C, Cronje H, Gonnet JM, Guillot M, Maria B, Moodley J, Oury JF, Thoulon JM, Treisser A, et al. Induction of labor with mifepristone (RU 486) in intrauterine fetal death. Am J Obstet Gynecol. 1990 Aug;163(2):540-2. doi: 10.1016/0002-9378(90)91193-g. PMID 2201190
- [Result] Urquhart DR, Templeton AA. The use of mifepristone prior to prostaglandin-induced mid-trimester abortion. Hum Reprod. 1990 Oct;5(7):883-6. doi: 10.1093/oxfordjournals.humrep.a137203. PMID 2266162
- [Result] Hofmeyr GJ, Gulmezoglu AM, Pileggi C. Vaginal misoprostol for cervical ripening and induction of labour. Cochrane Database Syst Rev. 2010 Oct 6;2010(10):CD000941. doi: 10.1002/14651858.CD000941.pub2. PMID 20927722
- [Result] Mariani Neto C, Leao EJ, Barreto EM, Kenj G, De Aquino MM, Tuffi VH. [Use of misoprostol for labor induction in stillbirth]. Rev Paul Med. 1987 Nov-Dec;105(6):325-8. No abstract available. Portuguese. PMID 3144030
- [Result] Bartha JL, Comino-Delgado R, Garcia-Benasach F, Martinez-Del-Fresno P, Moreno-Corral LJ. Oral misoprostol and intracervical dinoprostone for cervical ripening and labor induction: a randomized comparison. Obstet Gynecol. 2000 Sep;96(3):465-9. doi: 10.1016/s0029-7844(00)00954-6. PMID 10960643
- [Result] Titiz H, Wallace A, Voaklander DC. Manual removal of the placenta--a case control study. Aust N Z J Obstet Gynaecol. 2001 Feb;41(1):41-4. doi: 10.1111/j.1479-828x.2001.tb01292.x. PMID 11284645
- [Result] Gomez Ponce de Leon R, Wing D, Fiala C. Misoprostol for intrauterine fetal death. Int J Gynaecol Obstet. 2007 Dec;99 Suppl 2:S190-3. doi: 10.1016/j.ijgo.2007.09.010. Epub 2007 Oct 24. PMID 17961568
- [Result] Nicoll AE, Mackenzie F, Greer IA, Norman JE. Vaginal application of the nitric oxide donor isosorbide mononitrate for preinduction cervical ripening: a randomized controlled trial to determine effects on maternal and fetal hemodynamics. Am J Obstet Gynecol. 2001 Apr;184(5):958-64. doi: 10.1067/mob.2001.111797. PMID 11303205
- [Derived] Arteaga-Troncoso G, Chacon-Calderon AE, Martinez-Herrera FJ, Cruz-Nunez SG, Lopez-Hurtado M, Belmont-Gomez A, Guzman-Grenfell AM, Farfan-Labonne BE, Neri-Mendez CJ, Zea-Prado F, Guerra-Infante FM. A randomized controlled trial comparing isosorbide dinitrate-oxytocin versus misoprostol-oxytocin at management of foetal intrauterine death. PLoS One. 2019 Nov 21;14(11):e0215718. doi: 10.1371/journal.pone.0215718. eCollection 2019. PMID 31751343